CLINICAL TRIAL: NCT06155799
Title: Accuracy of Dynamic Navigation System on Zygomatic Implant Placement: A Randomized Clinical Trial
Brief Title: Accuracy of Dynamic Navigation System on Zygomatic Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Collaborators: Principal Investigator: Bassel Traboulsi-Garet. Master of Oral Surgery and Implantology. University of Barcelona (Unknown); Study Chair: Javier Bara-Casaus. Head of the Oral and Maxillofacial Surgery Institute. University Hospital Sagrat Cor, Barcelona. (Unknown); Study Chair: Eduard Valmaseda-Castellón. Full professor of Oral Surgery. University of Barcelona (Unknown); Study Chair: Octavi Camps-Font. Lecturer in Oral Surgery. University of Barcelona (Unknown); Study Director: Maria Angels Sanchez-Garces. Associate professor in Oral Surgery. University of Barcelona (Unknown)
Responsible Party: Principal Investigator, Adrià Jorba García, DDS, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/2023
Record Dates: First submitted 2023-11-21; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Dental Implants; Surgery, Computer-Assisted
Keywords: Surgery, Computer-Assisted; Dental implant; Navigation system

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patient will be unaware of which group since during the surgical procedure patient eyes' will be covered.
  Outcome assessor won't take part of the clinical process and will be blinded regarding which group is allocated each patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Navigation group (Experimental): Zygomatic implant placement by dynamic computer assisted surgery system.
  Interventions: Device: Freehand zygomatic implant placement
- Freehand group (Active Comparator): Zygomatic implant placement by Freehand, without any guidance.
  Interventions: Device: Freehand zygomatic implant placement

INTERVENTIONS:
Device: Freehand zygomatic implant placement — Zygomatic implants will be placed without any guidance after preoperative virtual planning has been performed.

SUMMARY:
This study consists in a randomized controlled trial which objective is to assess the accuracy of a dynamic navigation system in zygomatic implant placement in partially or total edentulous patients in the upper jaw compared with the conventional freehand method.

DETAILED DESCRIPTION:
The present study is a prospective randomized clinical trial.

Each patient enrolled in this trial will be randomly allocated to on group (Navigation group (test group) or Freehand group (control group)). Preoperative virtual planification of zygomatic an conventional implants on a prerequired cone beam computed tomography (CBCT) with radiographic markers (tooth if possible or micro implants if not possible) will be performed for each patient.

The patient will be randomly allocated in one group just before the surgery, and the surgical procedure will be performed according the surgery protocol of each group. Then, after the surgical procedure a PROMs questionnaire will be asked to the patients.

Finally a postoperative CBCT will be performed and overlapped with the preoperative CBCT with the implants planification and implant position deviations between the planned and final position will be measured.

The study devices are European Conformity (CE) marked products and used within their intended use.

ELIGIBILITY:
Inclusion Criteria:

* Partial or total edentulous maxilla
* Large bone atrophy that avoids possible conventional implant placement
* Over 18 years old patients

Exclusion Criteria:

* Patients with facial bone disease that contraindicates conventional or zygomatic implants placement.
* Systemic or local conditions that contraindicates oral surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Angular deviation | 1 month
  Angular deviation between the virtual planed position of the implant and the final implant position. Measured in degrees
Platform 3D deviation | 1 month
  Global deviation at the platform of the zygomatic implant between the virtual planned position and the final position of the dental implant measured in the 3 axes of the space (3D deviation). Measured in millimeters (mm).
Apex 3D deviation | 1 month
  Global deviation at the apex of the dental implant between the virtual planned position and the final position of the dental implant measured in the 3 axes of the space (3D deviation). Measured in millimeters (mm).

SECONDARY OUTCOMES:
Patient-reported outcome measures questionnaire | One week post operative
  Patients perception of therapy functional well-being and health status during the dental implant treatment with a navigation system. The scale goes from 0 to 4, where higher scores mean worse outcome.
Time of surgery | 24 hours
  Two times of surgery were recorded: time of drilling, from the first drilling of the first zygomatic implant to the last zygomatic implant placement; and time of complete surgery procedure, from first incision to suture.
Complications | 6 months
  Number of intra and postoperative complications and what kind of complication it was.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Odontológic de Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fan S, Saenz-Ravello G, Diaz L, Wu Y, Davo R, Wang F, Magic M, Al-Nawas B, Kammerer PW. The Accuracy of Zygomatic Implant Placement Assisted by Dynamic Computer-Aided Surgery: A Systematic Review and Meta-Analysis. J Clin Med. 2023 Aug 21;12(16):5418. doi: 10.3390/jcm12165418. PMID 37629460
- [Result] Kammerer PW, Fan S, Aparicio C, Bedrossian E, Davo R, Morton D, Raghoebar GM, Zarrine S, Al-Nawas B. Evaluation of surgical techniques in survival rate and complications of zygomatic implants for the rehabilitation of the atrophic edentulous maxilla: a systematic review. Int J Implant Dent. 2023 May 17;9(1):11. doi: 10.1186/s40729-023-00478-y. PMID 37198345
- [Result] Bhalerao A, Marimuthu M, Wahab A, Ayoub A. Dynamic navigation for zygomatic implant placement: A randomized clinical study comparing the flapless versus the conventional approach. J Dent. 2023 Mar;130:104436. doi: 10.1016/j.jdent.2023.104436. Epub 2023 Jan 31. PMID 36736529
- [Result] Tao BX, Wang F, Shen YH, Fan SQ, Huang W, Wang YP, Wu YQ. [Accuracy and clinical outcome of a real-time surgical navigation system for the placement of quad zygomatic implants]. Zhonghua Kou Qiang Yi Xue Za Zhi. 2020 Nov 9;55(11):845-850. doi: 10.3760/cma.j.cn112144-20200614-00343. Chinese. PMID 33171557
- [Result] Wu Y, Tao B, Lan K, Shen Y, Huang W, Wang F. Reliability and accuracy of dynamic navigation for zygomatic implant placement. Clin Oral Implants Res. 2022 Apr;33(4):362-376. doi: 10.1111/clr.13897. Epub 2022 Feb 15. PMID 35113463
- [Result] Tao B, Shen Y, Sun Y, Huang W, Wang F, Wu Y. Comparative accuracy of cone-beam CT and conventional multislice computed tomography for real-time navigation in zygomatic implant surgery. Clin Implant Dent Relat Res. 2020 Dec;22(6):747-755. doi: 10.1111/cid.12958. Epub 2020 Oct 28. PMID 33112508
- See also: Related Info — https://www.icmje.org/recommendations/browse/publishing-and-editorial-issues/clinical-trial-registration.html